CLINICAL TRIAL: NCT03115892
Title: The Effect of Mouthwash Containing Green Tea With Aloe Vera and Chlorhexidine Mouthwash on Oral Malodour Among a Group of Egyptian Children: Randomized Clinical Trial
Brief Title: Green Tea With Aloe Vera Mouthwash and Chlorohexidine Mouthwash
Acronym: RCT
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Asmaa Salah Eldin Abd El Samea Allam, oral and dental medicine , principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: pedodontics
Record Dates: First submitted 2017-04-12; First posted 2017-04-14 (Actual); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Halitosis
MeSH Terms: conditions — Halitosis | interventions — Tea

STUDY DESIGN:
Intervention Model Description: two group one for intervention and one for control randomize control trail
Masking Description: Statistician only will be blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention arm (Experimental): Green Tea With Aloe Vera mouthwash twice daily for one week
  Interventions: Drug: Green Tea With Aloe Vera mouthwash
- control arm (Active Comparator): Chlorhexidine Mouthwash twice daily for one week
  Interventions: Drug: Chlorhexidine mouthwash

INTERVENTIONS:
Drug: Green Tea With Aloe Vera mouthwash — measuring Tool/device Smell identification test ( organoleptic score ) (human nose) to measure of malodor which its unit 0-5 score
  Other Names: herbal mouthwash
  Arms: intervention arm
Drug: Chlorhexidine mouthwash — chlorohexidine mouthwash take two times per day for one week
  Other Names: Chemical mouthwash
  Arms: control arm

SUMMARY:
The Effect of Mouthwash Containing Green Tea With Aloe Vera and Chlorhexidine Mouthwash on Oral Malodour Among a Group of Egyptian Children: Randomized Clinical Trial

DETAILED DESCRIPTION:
1. Diagnosis:

1. Diagnostic chart (Appendix A) will be filled with personal, medical and dental history. DMF and def caries index (decayed, missing, and filled teeth).
2. The intra oral and extra oral examinations will be made using masks, gloves, cap, goggles, gauze, medical tray, dental mirror and WHO ( World Health Organization ) probe. All materials will be packaged in sterilizations wraps and autoclave, following the required bio safety standards

2. Intervention:

• The participants included will be allocated into two groups by drawing of sealed and opaque envelopes containing the codes "A" and "B".

Experimental Group:( intervention ) Green tea with Aloe- Vera

1. Preparation of green tea with aloe - Vera will occur under aseptic condition by pharmacist (Sargolzaie et al, 2015).
2. Collection of saliva samples (pre-rinse) will be obtained from children who fulfilled the inclusion criteria.
3. Distinguish odors using the Smell identification test (Doty et al. 1984). Breath was scored as described by Rosenberg at rest (open mouth without breathing) and when the patients counted from 1 to 11 (Rosenberg, 1996). A 0-5 score was given (Green man et al. 2004).
4. Subjects will be instructed to wash and retain the respective mouth rinse in the mouth for 40 Seconds before expectorating it.
5. 15 min after a rinse , Breath was scored as described by Rosenberg at rest (open mouth without breathing) and when the patients counted from 1 to 11 (Rosenberg, 1996). A 0-5 score was given (Green man et al. 2004). (masking effect)
6. Patients will not allow consuming any diet or drinking orally for following 90 min.
7. Again after 90 min, the saliva samples will be taken and inoculated on blood agar plates to determine the colony count (Velmurugan et al, 2013) and
8. Patients with confirmed oral malodor rinsed mouthwash during 7 days (15 ml, 2x/day for 1 min.)
9. After 7 days Breath was scored as described by Rosenberg at rest (open mouth without breathing) and when the patients counted from 1 to 11 (Rosenberg, 1996). A 0-5 score was given (Green man et al. 2004). (therapeutic effect).

Comparative Group:

Commercial Chlorhexidine 0.2%

1. Collection of saliva samples (pre-rinse) will be obtained from children who fulfilled the inclusion criteria.
2. Distinguish odors using the Smell identification test (Doty et al. 1984). Breath was scored as described by Rosenberg at rest (open mouth without breathing) and when the patients counted from 1 to 11 (Rosenberg, 1996). A 0-5 score was given (Green man et al. 2004).
3. Subjects will be instructed to wash and retain the respective mouth rinse in the mouth for 40 Seconds before expectorating it.
4. 15 min after a rinse , Breath was scored as described by Rosenberg at rest (open mouth without breathing) and when the patients counted from 1 to 11 (Rosenberg, 1996). A 0-5 score was given (Green man et al. 2004). (masking effect)
5. Patients will not allow consuming any diet or drinking orally for following 90 mins.
6. Again after 90 min, the saliva samples will be taken and inoculated on blood agar plates to determine the colony count (Velmurugan et al, 2013) .
7. Patients with confirmed oral malodor rinsed mouthwash during 7 days (15 ml, 2x/day for 1 min.)
8. After 7 days Breath was scored as described by Rosenberg at rest (open mouth without breathing) and when the patients counted from 1 to 11 (Rosenberg, 1996). A 0-5 score was given (Green man et al. 2004). (therapeutic effect).

ELIGIBILITY:
Inclusion Criteria:

* 1. Children aged between 6 and 12 years. 2. Children having normal occlusion, non-compromised oral health (brushed their teeth once-daily) using toothbrush and non-fluoridated toothpaste. And practicing no other oral hygiene measures.

Exclusion Criteria:

* 1. History of current or recent (at least for the past 1 month) antibiotic usage or other medications.

  2. Abscess, draining sinus, cellulitis, or other conditions requiring emergency dental treatment.

  3. Children with known history of allergy to any mouthrinse or drug. 4. Children who wore fixed or removable orthodontic appliances.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 27 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-09-01 (Estimated); Study Completion 2017-12-01 (Estimated)

PRIMARY OUTCOMES:
Oral malodor | one week
  Smell identification test (organoleptic ) (human nose)

SECONDARY OUTCOMES:
Streptococcal count | one week
  measuring Tool by using blood agar plate unit CFU/ml colony-forming units

CONTACTS AND LOCATIONS:
Overall Officials: sherif B eltweel, ass.prof, Study Director — cairo unversity
Locations (1):
- Oral An Dental Medicine Faculty, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
it will be available after finished

REFERENCES:
- [Result] Dadamio J, Van Tournout M, Teughels W, Dekeyser C, Coucke W, Quirynen M. Efficacy of different mouthrinse formulations in reducing oral malodour: a randomized clinical trial. J Clin Periodontol. 2013 May;40(5):505-13. doi: 10.1111/jcpe.12090. Epub 2013 Mar 13. PMID 23489103
- See also: paper — https://www.ncbi.nlm.nih.gov/pubmed/23489103?tool=bestpractice.bmj.com